CLINICAL TRIAL: NCT05198453
Title: The Impact of Vaccination in a Cohort of Patients Hospitalized for Acute COVID-19
Brief Title: Impact of Vaccination in Acute COVID-19
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Daša Stupica, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: Breakthrough covid
Record Dates: First submitted 2022-01-18; First posted 2022-01-20 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Vaccination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vaccinated patients with COVID-19
  Interventions: Biological: vaccination
- unvaccinated patients with COVID-19

INTERVENTIONS:
Biological: vaccination — patients who received COVID-19 vaccine
  Groups: vaccinated patients with COVID-19

SUMMARY:
The aim of this study was to evaluate the association between vaccination with one of the four SARS-CoV-2 vaccines authorized for use in the European Union-BNT162b2, ChAdOx-1S, mRNA-1273 or Ad.26.COV2.S-and progression to critically severe disease among adult patients with PCR-confirmed acute COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* age 18 yers or more
* hospitalized for acute COVID-19
* PCR confirmed infection with SARS-CoV-2

Exclusion Criteria:

* hospitalized for other conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
number (%) with critically severe disease | assessment performed at a minimum 30 days after admission

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
After a reasonable request.